CLINICAL TRIAL: NCT00392587
Title: A Randomised, Double-blind, Placebo-controlled Parallel Study to Assess the Safety, Tolerability,Pharmacodynamics and Steady State Pharmacokinetics of Repeated Doses of GW856553 in Patients With COPD
Brief Title: A Study To Investigate The Effects Of GW856553 On Patients With COPD (Chronic Obstructive Pulmonary Disease)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKI106209
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Pharmacodynamics; Pharmacokinetics; Tolerability; COPD; Safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW856553

SUMMARY:
The purpose of this study is to assess the safety of GW856553 in COPD patients and to assess its affects on their COPD disease after 14 days.

ELIGIBILITY:
Inclusion criteria:

* Women of childbearing potential
* Established history of COPD
* Cigarette smoking history greater than 10 pack years
* FEV1 between 40 and 80% of predicted normal for height, age and sex.

Exclusion criteria:

* Morbidly obese patients (body mass index >40)
* Hospitalisation or treatment for worsening of COPD in past 6 weeks
* History of increased liver function tests
* hypersensitivity to salbutamol or ipratropium bromide
* Blood pressure > 155/95

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08

PRIMARY OUTCOMES:
Measurements of adverse events, changes in heart rate, blood pressure, blood tests, heart function and lung function throughout the 14 day study. Exacerbations of COPD over the 14 day study. | 14 days

SECONDARY OUTCOMES:
Inhibition of inflammatory agents in the blood after 7 and 14 days of dosing. | after 7 and 14 days of dosing
Concentration of the drug in the blood after 1, 3, 7, 10 and 14 days of dosing. | after 1, 3, 7, 10 and 14 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin

REFERENCES:
- [Derived] Yang S, Lukey P, Beerahee M, Hoke F. Population pharmacokinetics of losmapimod in healthy subjects and patients with rheumatoid arthritis and chronic obstructive pulmonary diseases. Clin Pharmacokinet. 2013 Mar;52(3):187-98. doi: 10.1007/s40262-012-0025-6. PMID 23254770